CLINICAL TRIAL: NCT06140784
Title: A Three-Month Clinical Study to Assess the Gingivitis and Plaque Effects of Various Dentifrices
Brief Title: A Clinical Study to Assess the Gingivitis and Plaque Effects of Various Dentifrices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023043
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.76% Sodium Monofluorophosphate Dentifrice (Sham Comparator)
  Interventions: Drug: 0.76% Sodium Monofluorophosphate Dentifrice
- Marketed 0.454% Stannous Fluoride plus Arginine Dentifrice (Active Comparator)
  Interventions: Drug: 0.454% Stannous Fluoride Dentifrice
- Marketed 0.454% Stannous Fluoride Dentifrice (Active Comparator)
  Interventions: Drug: 0.454% Stannous Fluoride Dentifrice
- 0.454% Stannous Fluoride Dentifrice (Active Comparator)
  Interventions: Drug: 0.454% Stannous Fluoride Dentifrice

INTERVENTIONS:
Drug: 0.76% Sodium Monofluorophosphate Dentifrice — Whole mouth brushing with a toothpaste, twice daily for the duration of the study.
  Arms: 0.76% Sodium Monofluorophosphate Dentifrice
Drug: 0.454% Stannous Fluoride Dentifrice — Whole mouth brushing with a toothpaste, twice daily for the duration of the study.
  Arms: Marketed 0.454% Stannous Fluoride plus Arginine Dentifrice
Drug: 0.454% Stannous Fluoride Dentifrice — Whole mouth brushing with a toothpaste, twice daily for the duration of the study.
  Arms: Marketed 0.454% Stannous Fluoride Dentifrice
Drug: 0.454% Stannous Fluoride Dentifrice — Whole mouth brushing with a toothpaste, twice daily for the duration of the study.
  Arms: 0.454% Stannous Fluoride Dentifrice

SUMMARY:
The primary objective of this study is to evaluate the effect four different dentifrices have on gingivitis after 12 weeks of product use. The secondary objectives are to assess the effect four dentifrices, have on plaque and oral microbiome composition.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be in general good health as determined by the Investigator based on a review of the health history/update for participation in the trial;
* Have at least 16 gradable teeth;
* Have mild to moderate gingivitis with at least 20 bleeding sites;
* Agree to return for scheduled visits and follow the study procedures;
* Agree to refrain from use of any non-study oral hygiene products for the duration of the study;
* Agree to delay any elective dentistry, including dental prophylaxis, until the completion of the study;
* Agree to refrain from any oral hygiene the morning of your visit
* Agree to refrain from eating, drinking (except water), using tobacco, floss, use toothpicks, breath mints, or chew gum after performing your evening brushing.

Exclusion Criteria:

* Having taken antibiotic, anti-inflammatory, or anti-coagulant medications within 4 weeks of the Baseline Visit;
* Have any oral conditions that could interfere with study compliance and/or examination procedures, such as widespread caries, soft or hard tissue tumor of the oral cavity, or advanced periodontal disease;
* Having had a dental prophylaxis within 2 weeks of plaque sampling visits;
* Removable oral appliances;
* Fixed facial or lingual orthodontic appliances;
* Self-reported pregnancy or lactation;
* Any diseases or condition that might interfere with the safe participation in the study; and
* Inability to undergo study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2023-09-02 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Löe-Silness Gingivitis Evaluation | 3 Months
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).

SECONDARY OUTCOMES:
Löe-Silness Gingivitis Evaluation | Baseline
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).
Löe-Silness Gingivitis Evaluation | 1 Month
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).
Mean Turesky Modified Quigley-Hein Index | Baseline
  The Turesky Modified Quigley-Hein Index was scored on six surfaces (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual and mesiolingual) to assess plaque on all gradable teeth. Whole mouth average plaque scores were calculated for each subject and tooth surfaces by totaling the scores and dividing by the number of gradable sites examined. the scoring criteria is below; (0) No Plaque; (1) Separate flecks of plaque at the cervical margin; (2) A thin, continuous band of plaque (up to 1 mm) at the cervical margin; (3) A band of plaque wider than 1 mm, but covering less than one third of the side of the crown of the tooth; (4) Plaque covering at least one third, but less than two thirds of the side of the crown of the tooth; (5) Plaque covering two thirds or more of the side of the crown of the tooth.
Mean Turesky Modified Quigley-Hein Index | 1 Month
  The Turesky Modified Quigley-Hein Index was scored on six surfaces (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual and mesiolingual) to assess plaque on all gradable teeth. Whole mouth average plaque scores were calculated for each subject and tooth surfaces by totaling the scores and dividing by the number of gradable sites examined. the scoring criteria is below; (0) No Plaque; (1) Separate flecks of plaque at the cervical margin; (2) A thin, continuous band of plaque (up to 1 mm) at the cervical margin; (3) A band of plaque wider than 1 mm, but covering less than one third of the side of the crown of the tooth; (4) Plaque covering at least one third, but less than two thirds of the side of the crown of the tooth; (5) Plaque covering two thirds or more of the side of the crown of the tooth.
Mean Turesky Modified Quigley-Hein Index | 3 Months
  The Turesky Modified Quigley-Hein Index was scored on six surfaces (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual and mesiolingual) to assess plaque on all gradable teeth. Whole mouth average plaque scores were calculated for each subject and tooth surfaces by totaling the scores and dividing by the number of gradable sites examined. the scoring criteria is below; (0) No Plaque; (1) Separate flecks of plaque at the cervical margin; (2) A thin, continuous band of plaque (up to 1 mm) at the cervical margin; (3) A band of plaque wider than 1 mm, but covering less than one third of the side of the crown of the tooth; (4) Plaque covering at least one third, but less than two thirds of the side of the crown of the tooth; (5) Plaque covering two thirds or more of the side of the crown of the tooth.

CONTACTS AND LOCATIONS:
Locations (1):
- UHRG, Whittier, California, United States